CLINICAL TRIAL: NCT00767130
Title: DNA Diagnostic System for Statin Safety and Efficacy
Acronym: SIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genomas, Inc (Industry)
Collaborators: Hartford Hospital (Other); University of California, San Francisco (Other); Cornell University (Other)
Responsible Party: Gualberto Ruano/President, Genomas, Inc.
Other Study IDs: 1 R44 HL091697-01
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Hypercholesterolemia; Myopathy
Keywords: single nucleotide polymorphisms, SNP, LDL cholesterol, statin myopathy, atorvastatin, simvastatin, rosuvastatin
MeSH Terms: conditions — Hypercholesterolemia; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: receiving atorvastatin
- 2: receiving simvastatin
- 3: receiving rosuvastatin

SUMMARY:
Lipitor®, Zocor®, and Crestor® are statin drugs commonly taken to lower cholesterol and prevent heart disease. Statins lower cholesterol by different amounts in different patients and sometimes statins cause muscle pain, cramps, or weakness. This study will examine genetic differences in the blood of patients taking statins to predict both how well the statins lower cholesterol, and whether muscle discomfort occurs. Finding such genetic connections is the key to developing genetic tests that might eventually help determine which statin is best for a patient. About 1000 people will be in the study.

DETAILED DESCRIPTION:
Statin efficacy in primary and secondary prevention of cardiovascular disease has led to increasingly aggressive usage and dosage of statins. Their main clinically relevant safety risk is statin-induced myopathy (SIM) evidenced as a constellation of neuromuscular side effects (NMSE) that include myalgias (muscle aches, cramps, weakness) and myositis (monitored by elevation of serum creatine kinase [CK] activity). NMSEs are disabling to 3-20% of patients on statins, require alteration of therapy, and reduce compliance. NMSEs vary in extent between drugs and from patient to patient. We will develop a novel product termed SIM PhyzioType™ system to provide clinicians with individualized information for each patient on the safest statin drug among atorvastatin, simvastatin, and rosuvastatin, the 3 most prescribed statins. The PhyzioType consists of a multi-SNP (single nucleotide polymorphism) ensemble that, interpreted with a biomathematical algorithm, predicts drug response. We have developed a prototype PhyzioType system incorporating predictive models for myalgia, serum CK activity, and LDLc reduction for atorvastatin and simvastatin patients. We will recruit to obtain 250 patients treated with each drug and use existing clinical records to characterize their NMSE and LDLc responses. We will use physiogenomic analysis to identify those SNPs that differentiate the risk of NMSEs among the 3 statins and combine them into the SIM PhyzioType system. This work will also contribute to the pharmacology of SIM and unravel new pharmaceutical targets. We will create and validate the SIM PhyzioType system with clinically useful prediction of NMSEs and potency for each of the 3 statins. In Phase III a prospective trial is planned for FDA approval of the SIM PhyzioType product.

ELIGIBILITY:
Inclusion Criteria:

* receiving, or documented to have received in the past, any of the statins including atorvastatin, simvastatin, rosuvastatin treatment for hypercholesterolemia
* chart-documented clinical record of having had, never having had, or possibly having had, statin-associated myopathy

Exclusion Criteria:

* never having taken any statin medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated for hypercholesterolemia at Hartford Hospital, University of California-San Francisco, or the Rogosin Clinic at New York Presbyterian Hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
myopathy | in response to statin therapy
serum creatine kinase activity | in response to statin therapy

SECONDARY OUTCOMES:
LDL cholesterol | in response to statin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Ruano, MD, PhD, Principal Investigator — Genomas, Inc
Locations (3):
- United States (3):
  - University of California-San Francisco, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Rogosin Institute, New York Presbyterian Hospital, New York, New York

REFERENCES:
- [Background] Ruano G, Thompson PD, Windemuth A, Seip RL, Dande A, Sorokin A, Kocherla M, Smith A, Holford TR, Wu AH. Physiogenomic association of statin-related myalgia to serotonin receptors. Muscle Nerve. 2007 Sep;36(3):329-35. doi: 10.1002/mus.20871. PMID 17600820
- [Background] Ruano G, Thompson PD, Windemuth A, Smith A, Kocherla M, Holford TR, Seip R, Wu AH. Physiogenomic analysis links serum creatine kinase activities during statin therapy to vascular smooth muscle homeostasis. Pharmacogenomics. 2005 Dec;6(8):865-72. doi: 10.2217/14622416.6.8.865. PMID 16296949
- [Derived] Ruano G, Seip R, Windemuth A, Wu AH, Thompson PD. Laboratory Medicine in the Clinical Decision Support for Treatment of Hypercholesterolemia: Pharmacogenetics of Statins. Clin Lab Med. 2016 Sep;36(3):473-91. doi: 10.1016/j.cll.2016.05.010. Epub 2016 Jun 24. PMID 27514463
- [Derived] Ruano G, Windemuth A, Wu AH, Kane JP, Malloy MJ, Pullinger CR, Kocherla M, Bogaard K, Gordon BR, Holford TR, Gupta A, Seip RL, Thompson PD. Mechanisms of statin-induced myalgia assessed by physiogenomic associations. Atherosclerosis. 2011 Oct;218(2):451-6. doi: 10.1016/j.atherosclerosis.2011.07.007. Epub 2011 Jul 20. PMID 21868014
- See also: Hartford Hospital & the Henry Low Heart Center — http://www.harthosp.org/heart/default.aspx
- See also: Rogosin Institute, affiliated with NY Presbyterian Hospital and Weill Cornell School of Medicine — http://www.rogosin.org/index.php?id=36